CLINICAL TRIAL: NCT00228865
Title: Effects of Pulsatile IV Insulin on Cognitive Deficits in Diabetic Patients
Brief Title: Clinical Effects of Pulsatile Insulin Delivery on Cognitive Function- Phase 1
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Administrative
Sponsor: Florida Atlantic University (Other)
Collaborators: Advanced Diabetes Treatment Centers (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H09-66-COG
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes Mellitus
Keywords: Pulsatile intravenous insulin; Oral carbohydrate loading; Mindstream testing; Wechsler Memory Scale II; Respiratory Quotients; Hypoglycemia; Diabetes Mellitus with cognitive impairment; Diabetes Mellitus with complications
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia; Diabetes Complications | interventions — Insulin Aspart; Insulin, Regular, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Testing performed on diabetic patients with decline in cognitive function at baseline and quarterly after the start of receiving pulsatile intravenous insulin therapy to assess continuing cognitive function ability.
  Interventions: Procedure: Pulsatile IV insulin therapy; Procedure: Effects of Pulsatile IV Insulin on Cognitive functions

INTERVENTIONS:
Procedure: Pulsatile IV insulin therapy — Diabetic pts are given pulsatile iv insulin on a weekly basis determined by weekly phys orders based on pt response and insulin resistance. Cognitive testing is performed quarterly to track progress
  Other Names: Insulin includes Humulin, Humulog, Novolog and Epidra
Procedure: Effects of Pulsatile IV Insulin on Cognitive functions — Diabetic patients receive weekly treatment of Pulsatile Intravenous Insulin therapy. Dosage is determined each week by the patient's Endocrinologist based upon the patient's response and insulin resistance.
  Other Names: Humulin, Humulog

SUMMARY:
To determine if restoring normal metabolic function in patients with either Type I or Type II Diabetes can improve overall cognitive function. Patients are treated once a week with pulsatile intravenous insulin therapy mimicking normal insulin secretion and high amounts of oral glucose consumption.

DETAILED DESCRIPTION:
It is known that the glucose metabolic pathway (glycolysis) is the primary fuel generator in the brain and nerve tissue, the heart and vascular tissue, the eye, the kidney and the liver Deficient metabolic states such as seen in the glucose metabolism of diabetics can lead to sequelae. These damaging effects are exacerbated by altered cellular metabolites, specifically the increase in catabolic and decrease in anabolic factors. It has been shown over the past twenty years that normalization of metabolism in diabetic patients can be accomplished by mimicking the normal endogenous insulin pattern (ie., in pulses). Pulsatile insulin infusion has been demonstrated to reverse the diabetic metabolic state from primary fat utilization to carbohydrate utilization. This has been correlated with a stabilization of kidney function in patients with overt diabetic nephropathy, stabilization of blood glucoses, stabilization of blood pressure patterns, and reversal of hypoglycemic unawareness.

In patients with cognitive disorders (Alzheimer's type), infusion of intravenous insulin over a short interval (hours) improves cognitive function. Patients with this type of disorder have fewer insulin receptors in the affected areas of brain and insulin resistance by measurement of insulin and glucose levels in spinal fluid. This study is designed to study the effects of Pulsatile insulin on patients with diabetes mellitus and impaired cognitive function.

Diabetic individuals without other primary causes of cognitive impairment (brain tumor, previous neurosurgery, medications impairing memory) and able to swallow without difficulty will undergo pulsatile insulin treatments weekly over a period of 6-12 months with renewals for successive six month periods. Serial cognitive studies using Mindstream testing, Wechsler Memory Scale II and other localizing cognitive function tests will be done before the start of of treatment and every 3 months thereafter.This study began in 2002 and is continuing.

The respiratory quotient (RQ) is a measurement of CO2 exhaled and O2 inhaled and is proportionate to the fuel sources being used by the body, primarily the liver over short periods of time. The higher the RQ, the more glucose and less alternative fuel sources are being utilized. Following the RQ change helps determine the effectiveness of physiological insulin administration in increasing anabolic functions in diabetic individuals. By improving the body's glucose metabolism and thereby causing beneficial effects of anabolic factors, the possibility of serious complications can be decreased. In addition the use of oral carbohydrate at the same time along with the physiologic insulin administration stimulates the appropriate gut hormones which augment this effect, a response which cannot be duplicated with intravenous glucose. The purpose of our studies is to induce the physiologic administration of insulin along with the augmenting effect of oral carbohydrates, and by returning the normal fuel and organ metabolism as noted by RQ changes, evaluate its effectiveness in altering the deleterious effects on bodily functions in diabetic individuals.

The RQ is determined by the use of a metabolic cart. Individuals breathe into a mask for 3-5 minutes after a rest period of 30 or more minutes. The ratio of exhaled volume of CO2 to the inhaled volume of O2 is determined as the RQ. The physiologic range is 0.7 to1.3. Individuals using fat as a primary fuel have a ratio of 0.7, protein or mixed fuels is 0.8-0.9 and carbohydrate is 0.9-1.0. Those taking excessive calories will have RQ's higher than 1.05. The RQ can be followed serially and this is before and after each treatment. Three treatments are given during each visit to the center. The amount of intravenous insulin and oral glucose given is determined by the RQ changes during the previous treatment.

The treatment encourages the glucose metabolism in diabetics to normalize in multiple organs, especially muscle, retina, liver, kidney and nerve endings. The process fundamentally requires the administration of high dose insulin pulses similar to those found in non diabetic humans by their pancreas into the surrounding portal circulation. Oral carbohydrates are given simultaneously to augment the process and prevent hypoglycemia. The process is monitored by frequent glucose levels and respiratory quotients (RQ). RQ is measured by a metabolic cart which determines the ratio VCO2/ VO2. This ratio is specific for the fuel used at any one time by the body. The glucose levels are monitored to keep glucose levels appropriate and the RQ determines the need to readjust the infusion protocol in each patient for subsequent insulin infusion sessions.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:
* diagnosed with type 1 or type 2 diabetes mellitus.
* Self reporting or diagnosed with memory changes
* Taking oral agents and/or insulin for diabetic control
* Under Endocrinologist's supervision for diabetes management
* Endocrinologist must assess and approve patient for participation in this study
* Ability to swallow without difficulty
* Ability to commit to the weekly time requirements associated with the study

Exclusion Criteria:

* Other causes of cognitive impairment not related to diabetes
* Inability to take cognitive testing
* Lack of intravenous access
* Pregnancy
* Alcohol abuse, drug addiction or the use of illegal drugs
* Positive HIV
* Inability to breathe into machine for respiratory quotients

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2003-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
By utilizing Mindstream testing and/or Wechsler Memory Scale II on a quarterly basis to track the patients' progress, we will evaluate and document the outcomes of providing Metabolic Activation Therapy over a twelve month period. Documentation will inc | Testing performed at baseline and quarterly to compare and analyze patient's results after receiving pulsatile intravenous insulin therapy
Utilizing the Wechsler Memory Scale II, Type II diabetic patients are tested on recall on a quarterly basis to track improvement in cognitive function. | Testing performed at baseline and quarterly to evaluate progress in cognitive functions
Using repetitive respiratory quotients, we will assess the success of the reversal of the abnormal underlying metabolism in diabetic patients from primarily fat metabolism to carbohydrate metabolism. | Testing performed at the beginning and end of each pulsatile intravenous insulin therapy session to determine the need to modify the amount of insulin given to the patient

CONTACTS AND LOCATIONS:
Overall Officials: Betty Tuller, Ph.D., Principal Investigator — Florida Atlantic University
Locations (1):
- Florida Atlantic University, Boca Raton, Florida, United States

REFERENCES:
- [Background] Hammond GS, Aoki TT. Measurement of health status in diabetic patients. Diabetes impact measurement scales. Diabetes Care. 1992 Apr;15(4):469-77. doi: 10.2337/diacare.15.4.469. PMID 1499460
- [Background] Stewart R, Liolitsa D. Type 2 diabetes mellitus, cognitive impairment and dementia. Diabet Med. 1999 Feb;16(2):93-112. doi: 10.1046/j.1464-5491.1999.00027.x. PMID 10229302
- [Background] Gregg EW, Yaffe K, Cauley JA, Rolka DB, Blackwell TL, Narayan KM, Cummings SR. Is diabetes associated with cognitive impairment and cognitive decline among older women? Study of Osteoporotic Fractures Research Group. Arch Intern Med. 2000 Jan 24;160(2):174-80. doi: 10.1001/archinte.160.2.174. PMID 10647755
- [Background] Steen E, Terry BM, Rivera EJ, Cannon JL, Neely TR, Tavares R, Xu XJ, Wands JR, de la Monte SM. Impaired insulin and insulin-like growth factor expression and signaling mechanisms in Alzheimer's disease--is this type 3 diabetes? J Alzheimers Dis. 2005 Feb;7(1):63-80. doi: 10.3233/jad-2005-7107. PMID 15750215
- [Background] Watson GS, Craft S. Modulation of memory by insulin and glucose: neuropsychological observations in Alzheimer's disease. Eur J Pharmacol. 2004 Apr 19;490(1-3):97-113. doi: 10.1016/j.ejphar.2004.02.048. PMID 15094077